CLINICAL TRIAL: NCT00029523
Title: A Randomized Clinical Study to Determine the Patient Benefit and Safety of Depocyt (Cytarabine Liposome Injection) for the Treatment of Neoplastic Meningitis
Brief Title: DepoCyt Therapy in Patients With Neoplastic Meningitis From Lymphoma or a Solid Tumor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKY0101-010
Record Dates: First submitted 2002-01-15; First posted 2002-01-16 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Meningeal Neoplasms
Keywords: neoplastic; meningitis; cerebrospinal fluid; CSF; meningeal; meninges; CNS; Leptomeningeal Neoplasms
MeSH Terms: conditions — Meningeal Neoplasms; Meningitis | interventions — Cytarabine

INTERVENTIONS:
Drug: Intrathecal (injected into the spinal fluid) DepoCyt
Drug: Intrathecal methotrexate
Drug: Intrathecal cytarabine (also known as ara-C)

SUMMARY:
The purpose of this study is to find out how well an experimental drug called DepoCyt works for neoplastic meningitis (cancer that has spread to the tissues around the brain and spinal cord). DepoCyt is a new slow-release form of the cancer drug called ara-C (cytarabine). Cytarabine has been used for many years to treat cancer.

ELIGIBILITY:
* Diagnosed (or previously diagnosed) with lymphoma or a solid tumor (not leukemia)
* Diagnosed with neoplastic meningitis
* If female, not pregnant and will not become pregnant while on-study
* No other experimental therapy within 21 days of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-04; Study Completion 2004-11

PRIMARY OUTCOMES:
Progression-free survival, defined as the time to neurological progression or death

SECONDARY OUTCOMES:
Time to neurological progression;
Survival (all-cause and meningeal disease-specific)
Frequency of improvement in pre-existing meningeal-disease related neurological deficits
Karnofsky Performance Scores (KPS)
Quality of life
Cytological response rate
Overall safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Tutuncu, MD, PhD, Study Director — Pacira Pharmaceuticals, Inc
Locations (23):
- United States (21):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - University of Southern California, Norris Cancer Center, Los Angeles, California
  - University of Colorado Hospital, Anschutz Cancer Pavilion, Denver, Colorado
  - Georgetown University Medical Center Hematology/Oncology, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory Clinic, Department of Neurosurgery, Atlanta, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Rush Cancer Institute, Chicago, Illinois
  - Loyola University Medical Center, Dept. of Hematology/Oncology, Maywood, Illinois
  - Beth Israel Deaconess Medical Center Dept. of Neurology, Boston, Massachusetts
  - Park Nicollet Institute, Oncology Research Program, Minneapolis, Minnesota
  - JFK Neuroscience Institute, Edison, New Jersey
  - Bowman Gray School of Medicine/Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina
  - Case Western Reserve University Hospital of Cleveland, Cleveland, Ohio
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah, Hunsman Cancer Institute, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
- Canada (2):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Toronto Sunnybrook Regional Cancer Center, Toronto, Ontario

REFERENCES:
- [Background] Glantz MJ, Jaeckle KA, Chamberlain MC, Phuphanich S, Recht L, Swinnen LJ, Maria B, LaFollette S, Schumann GB, Cole BF, Howell SB. A randomized controlled trial comparing intrathecal sustained-release cytarabine (DepoCyt) to intrathecal methotrexate in patients with neoplastic meningitis from solid tumors. Clin Cancer Res. 1999 Nov;5(11):3394-402. PMID 10589750
- [Background] Glantz MJ, LaFollette S, Jaeckle KA, Shapiro W, Swinnen L, Rozental JR, Phuphanich S, Rogers LR, Gutheil JC, Batchelor T, Lyter D, Chamberlain M, Maria BL, Schiffer C, Bashir R, Thomas D, Cowens W, Howell SB. Randomized trial of a slow-release versus a standard formulation of cytarabine for the intrathecal treatment of lymphomatous meningitis. J Clin Oncol. 1999 Oct;17(10):3110-6. doi: 10.1200/JCO.1999.17.10.3110. PMID 10506606